CLINICAL TRIAL: NCT06173271
Title: The Effect of a Multi-intervention Program and Protein Food Sources on Preventing and Mitigating Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CMUH111-REC2-164
Record Dates: First submitted 2023-02-07; First posted 2023-12-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Dietary Exposure; Nutrition, Healthy; Bone Health; Muscle Function; Muscle Performance
Keywords: sarcopenia; protein; exercise; nutritional education; bone health
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Exercise only (Other): Exercise only (60 min/times, 3 times/wk)
  Interventions: Dietary Supplement: multi-intervention program and protein foods supplementation
- plant protein group (Active Comparator): Soymilk (230ml) and sweet potato (60g) supplementation after exercise (3 times/wk) plus nutrition education (once a wk)
  Interventions: Dietary Supplement: multi-intervention program and protein foods supplementation
- animal protein group (Active Comparator): Milk (240ml) and sweet potato (60g) supplementation after exercise (3 times/wk) plus nutrition education (once a wk)
  Interventions: Dietary Supplement: multi-intervention program and protein foods supplementation
- Control (No Intervention): No exercise and no nutrition education intervention
- Exercise and Nutrition Education group (Active Comparator): Exercise 60 min/times and three times per week Nutrition education 30 min/week
  Interventions: Dietary Supplement: multi-intervention program and protein foods supplementation

INTERVENTIONS:
Dietary Supplement: multi-intervention program and protein foods supplementation — This study aimed to investigate the effects of a multi-intervention program (protein-rich food supplement, nutrition education, and exercise) on reducing the risk of sarcopenia.
  Arms: Exercise and Nutrition Education group; Exercise only; animal protein group; plant protein group

SUMMARY:
Sarcopenia is characterized by loss of skeletal muscle mass and strength with advancing age. It is linked to an increased risk of falls, disability, length of hospitalization, poor quality of life, and burden of health care. Nutrition and physical activity are the major modifiable factors to prevent and mitigate sarcopenia. However, most studies focused on the explore the effects of physical activity or single nutrient supplementation. Whether a multi-intervention program combining protein-rich food intake, nutrition education, and exercise can more effectively reduce the risk of sarcopenia still needs to be explored at the community level. This study aimed to investigate the effects of a multi-intervention program (protein-rich food supplement, nutrition education, and exercise) on reducing the risk of sarcopenia. The primary outcome is to evaluate the effect of a multi-intervention program and exercise intervention only. The second outcome is to assess the impact of animal and plant source protein on muscle mass and physical performance. Investigators will recruit the study participants over the age of 60 from the free-living community. All participants were randomized into five groups: animal protein, plant protein, exercise and nutrition education, exercise alone, and control. For 8 weeks, except for control group, all four groups receive resistance training 3 times/week. However, the animal and plant protein groups provide milk 240 mL and soy milk 230 mL (7-8 g protein/serving) after exercise, respectively, and receive personal nutritional counseling and education to adhere to dietary recommendations. Dual-energy X-Ray using to evaluate the body composition and measure the grip strength, five-time chair stand test, and gait speed to assess physical performance pre- and post-intervention. The results of this study can be used to prevent muscle mass loss and frailty for older adults in the community.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 60 from the free-living community

Exclusion Criteria:

* Kidney patients, diabetics, cancer patients, moderate/severe cognitively impaired, disability, those who take any commercial protein nutritional supplements, those who are underweight, vegans, food allergy to dairy products and soy products

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The effect of a multi-intervention program and exercise intervention on muscle mass | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in muscle mass will be assessed by DXA in kilogram/meter2.
The effect of a multi-intervention program and exercise intervention on calf circumference | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in calf circumference will be assessed by tape in cm
The effect of a multi-intervention program and exercise intervention on grip strength | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in grip strength will be assessed by grip meter in kg
The effect of a multi-intervention program and exercise intervention on walking speed | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in walking speed will be assessed by timer in meters/second
The effect of a multi-intervention program and exercise intervention on sit-to-stand speed | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in sit-to-stand test will be assessed by timer in second

SECONDARY OUTCOMES:
The effect of a multi-intervention program and exercise intervention on dietary intake | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in dietary intake at 8 weeks will be assessed by questionnaire.

OTHER OUTCOMES:
The effect of a multi-intervention program and exercise intervention on bone density | From the date of the first time to collect the baseline data until the date of completion of the study (after intervention), assessed up to 12 weeks
  The changes from baseline in bone density will be assessed by DXA in T-score.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Huang, PhD, Principal Investigator — China Medical University, China
Locations (1):
- Yi-Chen Huang, Taichung, Baseline and Post Test of Intervention, Taiwan

REFERENCES:
- [Derived] Liao T, Wang TY, Lu MC, Kuo HL, Chen YL, Lin KC, Chen YL, Hsiao Y, Huang YC. Muscle performance and bone density following a multi-intervention program with milk or soy milk supplementation in older adults: quasi-experimental study. J Nutr Health Aging. 2026 Jan 22;30(3):100784. doi: 10.1016/j.jnha.2026.100784. Online ahead of print. PMID 41576679